CLINICAL TRIAL: NCT02771938
Title: Primary Radiotherapy And DIEP flAp Reconstruction Trial
Acronym: PRADA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR4328
Record Dates: First submitted 2016-05-11; First posted 2016-05-13 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
Keywords: radiotherapy, breast cancer, DIEP flap
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiotherapy before surgery (Experimental): Radiotherapy followed by mastectomy and DIEP flap reconstruction
  Interventions: Other: Radiotherapy before surgery

INTERVENTIONS:
Other: Radiotherapy before surgery — Radiotherapy followed by mastectomy and DIEP flap reconstruction

SUMMARY:
Many women with breast cancer now live for decades after their breast cancer treatment. In view of this, modern breast reconstruction surgery after mastectomy for breast cancer aims to reproduce as natural a breast shape as possible. Keeping a natural breast appearance has been shown to be very important to a woman's emotional and psychological recovery.

Breast cancer treatment often includes a combination of surgery, chemotherapy, radiotherapy, anticancer tablets such as Tamoxifen, and newer targeted drugs such as Herceptin. Radiotherapy is usually given after surgery. However, radiotherapy after mastectomy and breast reconstruction can damage the 'new' breast giving a less good breast shape and appearance in the longer term. Also, if recovery is slow following surgery, the radiotherapy is delayed which may reduce its effectiveness. Changing the order of treatments has been shown to be safe and effective for chemotherapy, Herceptin and anticancer tablets but we have very little information on giving radiotherapy before breast cancer surgery.

The investigators want to find out if giving radiotherapy before mastectomy and reconstruction alters surgical complication rates and they want to evaluate the appearance of the reconstructed breast when radiotherapy is given before surgery.

DETAILED DESCRIPTION:
Cancer outcomes are equivalent regardless of the order of systemic treatments and surgery with a trend towards improved overall survival in women age <50 years receiving chemotherapy before surgery. Adjuvant post-mastectomy chest wall RT has been shown to have both a local and survival benefit particularly in high risk patients. Accordingly, patients with T3/T4 breast cancer and/or with a significant burden of axillary disease commonly now receive a treatment sequence comprising primary chemotherapy followed by mastectomy and immediate autologous reconstruction, increasingly using abdominal fat (DIEP reconstruction), and finally adjuvant radiotherapy to the affected chest wall +/- supraclavicular fossa.

There are precedents for the use of upfront (neoadjuvant) radiotherapy (NART) followed by complex cancer surgery. For example, in rectal cancer, there is substantial evidence for the use of neoadjuvant chemotherapy and radiotherapy followed by aggressive surgical excision as the standard of care in patients with a threatened or involved circumferential margin. Short-course preoperative radiotherapy has been tested in multiple trials in rectal cancer, including the Swedish Rectal Cancer Trial, Dutch Colorectal Cancer Group Study and more recently the Medical Research Council CR07 trial. All three studies demonstrated better local control and improved disease-free and overall survival. Flap reconstruction of the perineum at the time of abdomino-perineal resection is well described as a method to reduce perineal morbidity and is indicated when primary closure cannot be achieved after wide local resection. By transferring a bulk of vascularized soft tissue into the irradiated pelvis, flap reconstruction has been shown to reduce infection rates, fill pelvic dead space, prevent wound dehiscence, and reduce time to healing. 'Short course' pre-operative rectal radiotherapy: surgery is generally undertaken 7-10 days after completion of radiotherapy with an acceptable impact on post-operative complication rate.

There is one published series of NART in breast cancer reporting an acceptable post-operative complication rate. Following on from this, surgeons and clinical oncologists from Imperial College and the Royal Marsden have begun to develop a limited experience of mastectomy and DIEP reconstruction 2-6 weeks following completion of radiotherapy (10 cases, no significant post-operative complications). This non-randomised phase I study sets out to formally evaluate the safety of reversing the order of mastectomy plus immediate DIEP flap reconstruction and adjuvant radiotherapy, with a view to a subsequent randomised controlled trial testing local control and cosmetic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women >18 years with histopathologically-confirmed breast cancer, who:
* require mastectomy for any reason (e.g. extensive disease, failed conservative management etc.)
* adjuvant radiotherapy and who are suitable for DIEP flap reconstruction at the time of mastectomy

Exclusion Criteria:

* Inability to give informed consent
* MDM unable to make recommendation for radiotherapy based on pre-operative histopathological and imaging findings ie mastectomy pathology required for MDM to decide on need/ target volume for post-mastectomy RT
* Severe chemotherapy toxicity affecting treatment planning schedule

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with presence of open breast wound | 4 weeks after mastectomy and DIEP flap reconstruction
  Presence of open breast wound at 4 weeks after mastectomy & DIEP flap reconstruction

SECONDARY OUTCOMES:
Volume and symmetry between the reconstructed and non-reconstructed breast using 3D-surface imaging | 3 months and 12 months after surgery
  Difference in volume and symmetry between the reconstructed and non-reconstructed breast using 3D-surface imaging at 3 months and 12 months after surgery.
Patient satisfaction | 3 months and 12 months after surgery
  Patient satisfaction (as measured using the BREAST-Q reconstruction module) before, three months after, and 12 months after surgery.
Applanation tonometry measure of breast compressibility between the reconstructed and non-reconstructed breast | 3 months and 12 months after surgery
  Difference in breast compressibility between the reconstructed and non-reconstructed breast using applanation tonometry at 3 months and 12 months following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona MacNeill, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thiruchelvam PTR, Leff DR, Godden AR, Cleator S, Wood SH, Kirby AM, Jallali N, Somaiah N, Hunter JE, Henry FP, Micha A, O'Connell RL, Mohammed K, Patani N, Tan MLH, Gujral D, Ross G, James SE, Khan AA, Rusby JE, Hadjiminas DJ, MacNeill FA; PRADA Trial Management Group. Primary radiotherapy and deep inferior epigastric perforator flap reconstruction for patients with breast cancer (PRADA): a multicentre, prospective, non-randomised, feasibility study. Lancet Oncol. 2022 May;23(5):682-690. doi: 10.1016/S1470-2045(22)00145-0. Epub 2022 Apr 7. PMID 35397804
- See also: Primary radiotherapy and deep inferior epigastric perforator flap reconstruction for patients with breast cancer (PRADA): a multicentre, prospective, non-randomised, feasibility study — https://doi.org/10.1016/S1470-2045(22)00145-0